CLINICAL TRIAL: NCT03048734
Title: A Pilot Study : Nocturnal Hypertension and Nocturia in African American Men
Brief Title: Nocturnal Hypertension and Nocturia in African American Men
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00046856
Record Dates: First submitted 2016-12-16; First posted 2017-02-09 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group (1): Men with Nocturia ≥2.
- Group (2): Men with no nocturia (0-1).

SUMMARY:
This study to obtain pilot data on Nocturnal Hypertension and Nocturia. In Dr. Victor's current NIH grant (Cut Your Pressure Too: The LA Barbershop Blood Pressure Study) the results show that uncontrolled systolic hypertension is independent determinantal of nocturia in African American men.

We now went to pursue this correlation by designing a new NIH grant Proposal to determine whether replacing short acting with long acting drugs and dosing them at bed time rather than in the morning will:

A. Lower the systolic Blood pressure during sleep B. Improve Nocturia and results in better sleep quality. The results suggest that short acting hydrochlorothiazide may contribute to nocturia in some patients.

DETAILED DESCRIPTION:
AIMS AND SIGNIFICANCE OF PILOT DATA

Determine:

1. The feasibility of Southern California registry as an effective measure to recruit African American men to participate in a new research program.
2. If men will comply with the study procedures including Actigraphy and ambulatory blood pressure monitors.
3. The within subject coefficient of variation for repeated measures of nocturnal blood pressure by ambulatory blood pressure monitoring, vertical activity at night by Actigraphy monitors.
4. Whether the ambulatory Blood pressure itself affects the sleep pattern on Actigraphy.
5. Nocturnal systolic blood pressure and nocturnal vertical activity are higher in men with self-reported nocturia ≥2 at night than in men with no reported nocturia.

Purpose:

Obtain key pilot data to show feasibility and document the reproducibility of the proposed measurements.

ELIGIBILITY:
Inclusion Criteria:

* African American Men
* Age 35 to 79 year-old
* Able to give informed consent
* Pass the home sleep study
* Willing to wear the wrist Actigraphy monitor for 9 days continuously.
* Willing to wear ambulatory blood pressure monitoring (ABPM) for 48 hours twice during the 9 days of the study period.

Exclusion Criteria:

* Diabetes Mellitus
* Taking Prostate medication
* Symptoms of prostate disease or urinary urgency
* Sleep apnea

  1. A neck circumference greater than 17 inches
  2. Using Continuous Positive Airway Pressure (CPAP)
  3. History of a diagnosis of Sleep Apnea
  4. Apnea Hypopnea Index (AHI) > 15 per hour

Ages: 35 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit men between 35 and 79 years old who are able to give informed consent, and are willing to be contacted for future research. Protocol will be approved by our Institutional Review Board and informed written consent will be obtained from all subjects.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of events of Nocturia in relation to blood pressure. | 9 days
  will evaluate the patients with how many times they go to the bathroom and assess the relation with their nocturnal blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Victor, MD, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No